CLINICAL TRIAL: NCT03747068
Title: Preoperative Use of ANTI-Tumor Necrosis Factor Therapy in Ulcerative Colitis Patients Who Underwent Ileal Pouch-Anal Anastomosis (IPAA) is Not Associated With Histological Fibrosis
Brief Title: The Influence of Biologcal Treatment on the Short-Term Complications of Surgery in Patients With Inflematory Bowel Disease.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Eran Zittan, Director of IBD unit, HaEmek Medical Center, Israel
Other Study IDs: 09-0218-E
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Ulcerative Colitis; Anti TNF Therapy; Ileal Pouch Anal Anastomosis (IPAA)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- anti-TNF: UC patients treated with maintenance anti-TNF therapy who underwent IPAA surgery
  Interventions: Drug: Anti-TNF Drug
- CONTROL GROUP: UC patients who were not exposed to anti-TNF therapy

INTERVENTIONS:
Drug: Anti-TNF Drug
  Groups: anti-TNF

SUMMARY:
BACKGROUND: Previous studies of short-term surgical outcomes after preoperative exposure to anti-TNF therapy in ulcerative colitis (UC) patients who have undergone IPAA have been conflicting. We sought to determine whether preoperative exposure to anti-TNF therapy affects histological measures of fibrosis in the colorectum, which may be a potential factor in adverse anastomosis complications following IPAA surgery.

METHODS: Individuals who received infliximab as maintenance therapy and who received their last dose within 180 days of the first stage of IPAA were selected. The control group comprised UC patients who were not exposed to anti-TNF therapy, matched by age, sex, BMI, disease duration, albumin levels, and post-operative leak outcome. Hematoxylin and eosin- (H&E) and trichrome-stained slides from the most distal, well-oriented, full-thickness section of colorectum from each patient's total colectomy specimen were evaluated. Blinded assessment of the degree of fibrosis in the lamina propria, the submucosa, the submucosa immediately adjacent to the muscularis propria, and the subserosa was performed by a single observer using a semi-quantitative pictorial scale.

ELIGIBILITY:
Inclusion Criteria:

* all individuals with IBD who underwent IPAA from January 2002 to June 2013 were reviewed .

Exclusion Criteria:

* Patients with CD
* Patients without adequate clinical records documenting the 30-day postoperative clinical outcomes .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with IBD who underwent IPAA from January 2002 to June 2013 were reviewed. Patients with CD and those without adequate clinical records documenting the 30-day postoperative clinical outcomes were excluded
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-10-09 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2015-10-09 (Actual)

PRIMARY OUTCOMES:
to determine whether preoperative exposure to anti-TNF therapy affects histological measures of fibrosis in the rectum, as increased rectal fibrosis may be a potential factor in adverse anastomosis complications following IPAA surgery | all individuals with IBD who underwent IPAA from January 2002 to June 2013 were reviewed
  Assesment of the degree of fibrosis in the lamina propria, the subbmucosa, the submucosa immediately adjacent to the muscularis propria, and the subserosa was performed by a single observer using a semi-quantitative pictorial scale.